CLINICAL TRIAL: NCT02488174
Title: Prevention of Severe Acute Respiratory Failure in Patients With PROOFcheck - an Electronic Checklist to Prevent Organ Failure
Brief Title: Prevention of Severe Acute Respiratory Failure in Patients With PROOFCheck
Acronym: PROOFcheck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michelle Gong, Professor, Albert Einstein College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2015-4775; UH3HL125119 (NIH)
Record Dates: First submitted 2015-03-18; First posted 2015-07-02 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Respiratory Failure; Multiple Organ Failure
MeSH Terms: conditions — Respiratory Insufficiency; Multiple Organ Failure | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Standard Care (Active Comparator): The pre-intervention control condition will be usual care: that is, clinicians practice as usual without clinician notification of risk and without prompting on care practices as recommended by PROOFcheck.
  Interventions: Other: Standard Care
- PROOFcheck (Experimental): The intervention for this study will consist of 3 parts: 1) Education of clinicians on prevention of severe ARF and MOF in and out of the ICU, and best practice with regards to patients with severe ARF; 2) Clinicians will be notified that a patient they are taking care of has been identified as being at high risk for developing severe ARF requiring prolong MV; 3) Notified clinicians will be directed to PROOFcheck with a bundle of recommendations for best care for patients with ARF.
  Interventions: Other: PROOFcheck

INTERVENTIONS:
Other: PROOFcheck
  Arms: PROOFcheck
Other: Standard Care
  Arms: Standard Care

SUMMARY:
Severe acute respiratory failure (ARF) requiring prolonged mechanical ventilation is the most common form of acute organ dysfunction in the hospital, and is often associated with multiple organ failure (MOF), high mortality, and functional impairment. Most studies on ARF have focused on patients in the intensive care unit (ICU) after they have been on mechanical ventilation for days and end organ damage is already established. The overall goal of this proposed project is to improve the outcomes of patients at high risk for developing severe ARF and prolonged mechanical ventilation in and outside of the ICU. The project aims to intervene early in high risk patients with an electronic medical records (EMR)-based, patient-centered checklist of common critical care practices aimed at preventing lung injury and hospital acquired adverse events that commonly lead to organ failure (Prevention of Organ Failure checklist -PROOFcheck). This application proposes a stepped-wedge, clustered randomized control trial to determine the utility of PROOFcheck to improve survival and reduce the duration of mechanical ventilation and multiple organ failure in patients identified as high risk for progressing to severe ARF and prolonged mechanical ventilation. The aims in the UH2 phase are: 1) to refine a previously validated Lung Injury Prediction Score into a pragmatic, EMR-based early prediction model to Accurately Predict Prolonged Ventilation (APPROVE), which will automatically identify patients anywhere in the hospital who are at high risk for developing severe ARF requiring mechanical ventilation >48 hours; 2) to incorporate PROOFcheck into the EMR to prompt clinicians on care practices to limit lung injury, prevent adverse events, and avoid additional organ failure; and 3) to establish the infrastructure for the proposed trial. The proposed pragmatic trial will harness the hospital-wide EMR to identify patients at high risk for prolonged mechanical ventilation with APPROVE for intervention with PROOFcheck. As such, the proposed trial aims to break out of the clinical silos by which care is currently organized in the hospital and bring patient-centered, context appropriate care to the acutely ill patient wherever and whenever the patient's condition requires it.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged > 18 in the hospital
* Identified as being at high risk for developing severe ARF requiring prolonged MV

Exclusion Criteria:

* Patients who are chronically ventilated
* Patients who have DNI orders on hospital admission
* Patients in areas of the hospital that are unable or unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34040 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality | up to 1 year

SECONDARY OUTCOMES:
Hospital Length of Stay | up to 1 year
Organ Failure | up to 7 days
  SOFA score
Ventilator Free Days | up to 28 days
6 Month Mortality | up to 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- [Derived] Dziadzko MA, Novotny PJ, Sloan J, Gajic O, Herasevich V, Mirhaji P, Wu Y, Gong MN. Multicenter derivation and validation of an early warning score for acute respiratory failure or death in the hospital. Crit Care. 2018 Oct 30;22(1):286. doi: 10.1186/s13054-018-2194-7. PMID 30373653
- [Derived] Gong MN, Schenk L, Gajic O, Mirhaji P, Sloan J, Dong Y, Festic E, Herasevich V. Early intervention of patients at risk for acute respiratory failure and prolonged mechanical ventilation with a checklist aimed at the prevention of organ failure: protocol for a pragmatic stepped-wedged cluster trial of PROOFCheck. BMJ Open. 2016 Jun 10;6(6):e011347. doi: 10.1136/bmjopen-2016-011347. PMID 27288382